CLINICAL TRIAL: NCT03197324
Title: A Phase 1, Open-label, Randomized, Two-period, Two-treatment, Crossover Study to Evaluate the Effect of Bexagliflozin on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: Bexagliflozin Drug/Drug Interaction Study With Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-443
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — bexagliflozin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Digoxin Alone first, then Digoxin With Bexagliflozin (Active Comparator)
  Interventions: Drug: Digoxin
- Digoxin with Bexagliflozin, then Digoxin alone (Active Comparator)
  Interventions: Drug: Bexagliflozin; Drug: Digoxin

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablets, 20 mg
  Other Names: EGT0001442, EGT0001474
  Arms: Digoxin with Bexagliflozin, then Digoxin alone
Drug: Digoxin — 2 0.25 mg Digoxin tablets (total dose 0.5 mg digoxin)

SUMMARY:
The purpose of this study is to examine the drug-drug interaction in your body when given the study drug, bexagliflozin, with the heart failure medication digoxin. The study will evaluate whether bexagliflozin effects the amount of digoxin in your blood and how safe the study drug is and how well the study drug is tolerated when taken with digoxin.

DETAILED DESCRIPTION:
This was a phase 1, single center, open-label, two-period, two-treatment, crossover study to evaluate the effect of bexagliflozin tablets, 20 mg, on the pharmacokinetics (PK) of digoxin, 0.5 mg after co-administration in healthy subjects. Each subject was randomized into one of 2 treatment groups and participated in 2 treatment periods as outlined below. During the duration of the study, each subject received 8 single doses of bexagliflozin and 2 single doses of digoxin. Clinical laboratory tests and safety monitoring were conducted during Periods 1 and 2.

Group 1 - Period 1, Treatment A Subjects were admitted to the clinic on Day 0. Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, starting on Day 1 for 8 days, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 3. Blood samples for PK were drawn at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours (h) on Day 3, 24 h (Day 4), 48 h (Day 5), 72 h (Day 6), 96 h (Day 7), and 120 h (Day 8) after administration of digoxin. Subjects were discharged on Day 8.

Group 1 - Period 2, Treatment B Subjects were admitted to the clinic on Day 18. On Day 19, subjects received a single oral dose of 0.5 mg digoxin. Blood samples for PK were drawn at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 h on Day 19, 24 h (Day 20), 48 h (Day 21), 72 h (Day 22), 96 h (Day 23), and 120 h (Day 24) after administration of digoxin. Subjects were discharged on Day 24.

Group 2 - Period 1, Treatment B Subjects were admitted to the clinic on Day 0. On Day 1, subjects received a single oral dose of 0.5 mg digoxin. Blood samples for PK were drawn at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 h on Day 1, 24 h (Day 2), 48 h (Day 3), 72 h (Day 4), 96 h (Day 5), and 120 h (Day 6) after administration of digoxin. Subjects were discharged on Day 6.

Group 2 - Period 2, Treatment A Subjects were admitted to the clinic on Day 14. Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, for 8 days starting on Day 15, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 17. Blood samples for PK were drawn at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 h on Day 17, 24 h (Day 18), 48 h (Day 19), 72 h (Day 20), 96 h (Day 21), and 120 h (Day 22) after administration of digoxin. Subjects were discharged on Day 22.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2
2. Subjects who are non-smokers for at least 6 months prior to first dose
3. Subjects who are willing to use an adequate form of birth control during the study and for 30 days after discharge from clinic

Exclusion Criteria:

1. Subjects with a clinically significant history of allergy to drugs or latex
2. Subjects with a history of alcohol or drug dependence in the past 12 months
3. Subjects who have donated a significant amount of blood in the past 2 months
4. Subjects who have taken an investigational drug in the past 30 days or 7 half-lives of the investigational drug, whichever is longer
5. Subjects who had previously received digoxin or drugs of the same class, or SGLT2 inhibitors, in the past 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Director — Massachusetts General Hospital
Locations (1):
- Covance CRU, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this crossover study, the subject was to participate in 2 periods during which subjects received 2 treatments (A: Bexagliflozin co-administered with digoxin, B: Digoxin alone).
Groups:
- Digoxin and Bexagliflozin Tablet, Then Digoxin Alone: Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, starting on Day 1 for 8 days, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 3.
  Subjects were discharged on Day 8.
  On Day 19, subjects received a single oral dose of 0.5 mg digoxin and were discharged on Day 22.
- Digoxin, Then Digoxin and Bexagliflozin: On Day 1, subjects received a single oral dose of 0.5 mg digoxin. Subjects were discharged on Day 6.
  Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, for 8 days starting on Day 15, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 17. Subjects were discharged on Day 22.
Period: Overall Study
Arm/Group | Digoxin and Bexagliflozin Tablet, Then Digoxin Alone | Digoxin, Then Digoxin and Bexagliflozin
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes subjects dosed with any study drug.
Groups:
- Bexagliflozin and Digoxin, Then Digoxin Alone: Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, starting on Day 1 for 8 days, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 3
- Digoxin Alone, Then Bexagliflozin and Digoxin: On Day 1, subjects received a single oral dose of 0.5 mg digoxin. Subjects received daily oral doses of a bexagliflozin tablet, 20 mg, for 8 days starting on Day 15, and a single oral dose of 0.5 mg digoxin (two 0.25 mg tablets) was co-administered with bexagliflozin on Day 17.
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin and Digoxin, Then Digoxin Alone | Digoxin Alone, Then Bexagliflozin and Digoxin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (8.84) | 35.2 (6.37) | 40.0 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 73.6 (11.28) | 74.2 (13.67) | 73.9 (12.20)
Height [Mean (Standard Deviation); unit: cm] | 167.1 (8.44) | 165.6 (9.35) | 166.4 (8.71)

OUTCOME MEASURES:

1. Primary Outcome: Digoxin Cmax (Maximum Observed Plasma Concentration)
Description: Blood samples for pharmacokinetic parameters were drawn at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 h after administration of digoxin
Time Frame: Up to 120 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Digoxin Alone: Digoxin: Two 0.25 mg Digoxin tablets (total dose 0.5 mg digoxin)
- Digoxin With Bexagliflozin: Bexagliflozin: Bexagliflozin tablets, 20 mg
  Digoxin: Two 0.25 mg Digoxin tablets (total dose 0.5 mg digoxin)
Arm/Group | Digoxin Alone | Digoxin With Bexagliflozin
Number analyzed (Participants) | 20 | 19
ng/mL | 2.315 (28.8) | 2.301 (40.9)
Statistical Analysis 1: Comparison: Digoxin Alone vs Digoxin With Bexagliflozin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 100.40, 90% CI 2-sided [86.49 to 116.56] — Digoxin group is the denominator and Digoxin with Bexagliflozin is the numerator. Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subjects as a random effect

2. Primary Outcome: Digoxin Tmax (Time of Maximum Observed Plasma Concentration)
Description: as for outcome 1
Time Frame: Up to 120 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Digoxin Alone | Digoxin With Bexagliflozin
Number analyzed (Participants) | 20 | 19
hours | 1.00 [1 to 2] | 1.00 [1 to 4]

3. Primary Outcome: Digoxin T1/2 (Apparent Terminal Elimination Half-life)
Description: as for outcome 1
Time Frame: Up to 120 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Digoxin Alone | Digoxin With Bexagliflozin
Number analyzed (Participants) | 18 | 18
hours | 34.3 (15.5) | 38.2 (15.7)

4. Primary Outcome: AUC0-inf (Area Under the Plasma Concentration-time Curve From Time 0 to Infinity)
Description: as for outcome 1
Time Frame: Up to 120 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Digoxin Alone | Digoxin With Bexagliflozin
Number analyzed (Participants) | 18 | 18
h*ng/mL | 35.558 (16.6) | 37.805 (27.5)
Statistical Analysis 1: Comparison: Digoxin Alone vs Digoxin With Bexagliflozin; Geometric LS Mean was used as PK parameters; Test type: Superiority — Compare if co-administration of digoxin with bexagliflozin had significant impact on the PK of digoxin; Ratio of Geometric LSM = 106.12, 90% CI 2-sided [95.82 to 117.53] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 24 of the study
Arm/Group | Digoxin Alone | Digoxin With Bexagliflozin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 3/20 | 5/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin Alone (N=20) | Digoxin With Bexagliflozin (N=19)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI does not have the right to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03197324/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT03197324/SAP_001.pdf